CLINICAL TRIAL: NCT07145281
Title: Comparing the Effects of Sublingual Estradiol Treatment Versus Oral Estradiol With Cyproterone Acetate (CPA) Treatment on The Coagulation System in Transgender Women: A Prospective, Controlled Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Shmuel Kivity, MD, IRB Head, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0388-22-TLV; MOH_2022-10-11_012120 (Other: Israel Ministry of Health)
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria, Adult; Blood Coagulation; Coagulation Factors; Transgender Persons, M01.777.500; Hemostasis; Transgender Women
Keywords: Transgender women; sublingual estradiol; procoagulant effect; Protein S; Thrombin generation assay (TGA); Gender-affirming hormone therapy (GAHT)
MeSH Terms: conditions — Gender Dysphoria; Thrombosis | interventions — Estradiol; estradiol, estriol drug combination; Cyproterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual Estradiol (Experimental): Participants receive sublingual estradiol 2 mg per day divided into 4 doses, without an anti-androgen, for 6 months.
  Interventions: Drug: Estradiol (E2)
- Oral Estradiol + Cyproterone Acetate (CPA) (Active Comparator): Participants receive oral estradiol 2 mg once daily combined with cyproterone acetate 10 mg once daily for 6 months. This represents the standard regimen used in routine care.
  Interventions: Drug: Estradiol (E2); Drug: Cyproterone Acetate (Androcur, BAY94-8367)

INTERVENTIONS:
Drug: Estradiol (E2) — Participants receive estradiol 2 mg/day. In the experimental arm, estradiol is administered sublingually in four divided doses (0.5 mg each).
  In the active comparator arm, estradiol is administered orally, in combination with cyproterone acetate, for 6 months.
  All participants are treatment-naive.
  Other Names: Estrofem
Drug: Cyproterone Acetate (Androcur, BAY94-8367) — Participants in the active comparator arm receive cyproterone acetate (CPA) 10 mg orally, once daily, in combination with oral estradiol, for 6 months.
  All participants are treatment-naive.
  Arms: Oral Estradiol + Cyproterone Acetate (CPA)

SUMMARY:
The goal of this clinical trial is to learn about the effects of different routes of estradiol administration on blood clotting in transgender women starting gender-affirming hormone therapy. The main questions it aims to answer are:

Does sublingual estradiol reduce free Protein S levels compared to oral estradiol with cyproterone acetate?

Does sublingual estradiol accelerate activation of the clotting system, as measured by thrombin generation?

Researchers will compare sublingual estradiol to oral estradiol plus cyproterone acetate to see if the way estradiol is taken changes blood clotting risk.

Participants will:

Take either sublingual estradiol (2 mg daily in divided doses) or oral estradiol (2 mg daily) with cyproterone acetate (10 mg daily) for 6 months

Provide blood samples at baseline and after 6 months to measure hormone levels and clotting factors

Attend clinic visits for monitoring, including safety checks and routine laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* Self-identified transgender women
* Aged 18 to 45 years
* Healthy individuals
* Treatment-naïve (not previously exposed to gender-affirming hormone therapy)
* Presenting for gender-affirming hormone therapy (GAHT)
* Provided written informed consent

Exclusion Criteria:

* Active smokers
* Personal or family history of venous thromboembolism (VTE) or thrombophilia
* History of malignancy in the past 5 years
* Chronic liver disease
* Chronic kidney disease
* Hyperlipidemia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified transgender women (individuals assigned male at birth who identify as female) were eligible to participate in this study. Eligibility was limited to this gender identity.
Enrollment: 30 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Plasma Free Protein S Antigen Concentration at 6 Months | Baseline and 6 months after initiation of therapy
  Plasma concentration of free Protein S antigen will be measured at baseline and after 6 months of treatment. A reduction of ≥20% in free Protein S is anticipated in the sublingual estradiol group, with no comparable change expected in the oral estradiol group.

SECONDARY OUTCOMES:
Change in Protein C from baseline to 6 months | Baseline and 6 months after initiation of therapy
  Plasma concentration of Protein C antigen will be measured using immunologic assays at baseline and after 6 months of treatment.
Change in Prothrombin Time (PT) from baseline to 6 months | Baseline and 6 months after initiation of therapy
  PT will be measured at baseline and after 6 months using conventional clotting assays to evaluate changes in coagulation function.
Change from Baseline in Partial Thromboplastin Time (PTT) at 6 Months | Baseline and 6 months after initiation of therapy
  PTT will be measured at baseline and after 6 months using conventional clotting assays to evaluate changes in intrinsic coagulation pathway function
Change from Baseline in International Normalized Ratio (INR) at 6 Months | Baseline and 6 months after initiation of therapy
  INR will be measured at baseline and after 6 months using standard prothrombin time-based assays to assess changes in coagulation status.
Change from Baseline in Thromboelastography (TEG) Reaction Time (R Time) at 6 Months | Baseline and 6 months after initiation of therapy
  TEG Reaction Time (R time) will be measured at baseline and after 6 months using thromboelastography. R time is defined as the latency period from the start of the test until initial fibrin formation begins, reflecting the initiation phase of coagulation.
Change from Baseline in Thromboelastography (TEG) Maximum Amplitude (MA) at 6 Months | Baseline and 6 months after initiation of therapy
  TEG Maximum Amplitude (MA) will be measured at baseline and after 6 months using thromboelastography. MA reflects the maximum strength of the formed clot and is influenced by platelet function and fibrinogen levels.
Change from Baseline in Thrombin Generation Assay (TGA) Lag Time at 6 Months | Baseline and 6 months after initiation of therapy
  Lag time in the thrombin generation assay will be measured at baseline and after 6 months. TGA lag time represents the time until the initiation of thrombin generation, reflecting the onset of the coagulation process.
Change from Baseline in Thrombin Generation Assay (TGA) Peak Thrombin at 6 Months | Baseline and 6 months after initiation of therapy
  Peak thrombin levels will be measured using thrombin generation assay at baseline and after 6 months. This metric represents the highest concentration of thrombin generated during the assay and reflects the overall procoagulant potential.
Change from Baseline in Thrombin Generation Assay (TGA) Area Under the Curve (AUC) at 6 Months | Baseline and 6 months after initiation of therapy
  The area under the curve (AUC) in the thrombin generation assay will be calculated at baseline and after 6 months. AUC reflects the total amount of thrombin generated over time, providing a global measure of thrombin-generating capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Yaish, MD, Principal Investigator — Institute of Endocrinology, Metabolism and Hypertension, Tel Aviv Sourasky Medical Center, Tel Aviv
Locations (1):
- Tel Aviv Sourasky Medical Center - Institute of Endocrinology, Metabolism and Hypertension, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data (IPD), including baseline characteristics, hormonal and metabolic parameters, and hemostatic assay results collected during the 6-month intervention period, will be shared via the Open Science Framework repository (DOI: 10.17605/OSF.IO/TCRUW).
Time Frame: The individual participant data (IPD) set is already available and was uploaded to the Open Science Framework (OSF) repository. The data will remain accessible indefinitely unless otherwise specified in the repository.
Access Criteria: All researchers will be able to access the de-identified individual participant data (IPD) through the Open Science Framework (OSF) repository. The dataset includes baseline characteristics, laboratory results, and hemostatic parameters collected throughout the 6-month study period. Access is open and unrestricted via the following link: https://doi.org/10.17605/OSF.IO/TCRUW
  . No registration or approval process is required.
URL: https://doi.org/10.17605/OSF.IO/TCRUW

REFERENCES:
- [Background] Hembree WC, Cohen-Kettenis PT, Gooren L, Hannema SE, Meyer WJ, Murad MH, Rosenthal SM, Safer JD, Tangpricha V, T'Sjoen GG. Endocrine Treatment of Gender-Dysphoric/Gender-Incongruent Persons: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2017 Nov 1;102(11):3869-3903. doi: 10.1210/jc.2017-01658. PMID 28945902
- [Background] Dhejne C, Van Vlerken R, Heylens G, Arcelus J. Mental health and gender dysphoria: A review of the literature. Int Rev Psychiatry. 2016;28(1):44-57. doi: 10.3109/09540261.2015.1115753. PMID 26835611
- [Background] Ali-Saleh M, Sarig G, Ablin JN, Brenner B, Jacob G. Inhalation of a Short-Acting beta2-Adrenoreceptor Agonist Induces a Hypercoagulable State in Healthy Subjects. PLoS One. 2016 Jul 5;11(7):e0158652. doi: 10.1371/journal.pone.0158652. eCollection 2016. PMID 27379911
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders (5th ed.). Arlington, VA: American Psychiatric Association; 2013.
- [Background] Even Zohar N, Sofer Y, Yaish I, Serebro M, Tordjman K, Greenman Y. Low-Dose Cyproterone Acetate Treatment for Transgender Women. J Sex Med. 2021 Jul;18(7):1292-1298. doi: 10.1016/j.jsxm.2021.04.008. Epub 2021 Jun 24. PMID 34176757
- [Background] Connors JM, Middeldorp S. Transgender patients and the role of the coagulation clinician. J Thromb Haemost. 2019 Nov;17(11):1790-1797. doi: 10.1111/jth.14626. Epub 2019 Sep 13. PMID 31465627
- [Background] Dupuis M, Severin S, Noirrit-Esclassan E, Arnal JF, Payrastre B, Valera MC. Effects of Estrogens on Platelets and Megakaryocytes. Int J Mol Sci. 2019 Jun 25;20(12):3111. doi: 10.3390/ijms20123111. PMID 31242705
- [Background] Yokota N, Inoue R, Kawamura K, Egashira K, Kuma H, Kato K. The effects of dienogest and combined oral contraceptives on protein S-specific activity in endometriosis patients. Eur J Obstet Gynecol Reprod Biol. 2024 Apr;295:67-74. doi: 10.1016/j.ejogrb.2024.01.028. Epub 2024 Jan 29. PMID 38340593
- [Background] Mihaila RG, Catana C, Olteanu AL, Birlutiu V, Salcudean C, Mihaila MD. Thrombin generation is increased in patients with Clostridium difficile colitis - a pilot study. Biomarkers. 2019 Jun;24(4):389-393. doi: 10.1080/1354750X.2019.1600021. Epub 2019 Apr 9. PMID 30907672
- [Background] Volod O, Runge A. The TEG 5000 System: System Description and Protocol for Measurements. Methods Mol Biol. 2023;2663:725-733. doi: 10.1007/978-1-0716-3175-1_48. PMID 37204748
- [Background] Toorians AW, Thomassen MC, Zweegman S, Magdeleyns EJ, Tans G, Gooren LJ, Rosing J. Venous thrombosis and changes of hemostatic variables during cross-sex hormone treatment in transsexual people. J Clin Endocrinol Metab. 2003 Dec;88(12):5723-9. doi: 10.1210/jc.2003-030520. PMID 14671159
- [Background] van Ommen CH, Fijnvandraat K, Vulsma T, Delemarre-Van De Waal HA, Peters M. Acquired protein S deficiency caused by estrogen treatment of tall stature. J Pediatr. 1999 Oct;135(4):477-81. doi: 10.1016/s0022-3476(99)70171-x. PMID 10518082
- [Background] Raps M, Helmerhorst FM, Fleischer K, Dahm AE, Rosendaal FR, Rosing J, Reitsma P, Sandset PM, van Vliet HA. The effect of different hormonal contraceptives on plasma levels of free protein S and free TFPI. Thromb Haemost. 2013 Apr;109(4):606-13. doi: 10.1160/TH12-10-0771. Epub 2013 Feb 14. PMID 23407778
- [Background] Majumder R, Nguyen T. Protein S: function, regulation, and clinical perspectives. Curr Opin Hematol. 2021 Sep 1;28(5):339-344. doi: 10.1097/MOH.0000000000000663. PMID 34224431
- [Background] Bogehave M, Glintborg D, Christensen LL, T'Sjoen G, Vervalcke J, Wiepjes CM, den Heijer M, Andersen MS, Bladbjerg EM. The thrombin generation potential increases after feminizing gender-affirming hormone treatment, decreases after masculinizing gender-affirming hormone treatment, and is determined by the hormone treatment regimen. J Thromb Haemost. 2025 Oct;23(10):3084-3097. doi: 10.1016/j.jtha.2025.03.006. Epub 2025 Mar 14. PMID 40090622
- [Background] Lim HY, Leemaqz SY, Torkamani N, Grossmann M, Zajac JD, Nandurkar H, Ho P, Cheung AS. Global Coagulation Assays in Transgender Women on Oral and Transdermal Estradiol Therapy. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa262. doi: 10.1210/clinem/dgaa262. PMID 32413907
- [Background] Scheres LJJ, Selier NLD, Nota NM, van Diemen JJK, Cannegieter SC, den Heijer M. Effect of gender-affirming hormone use on coagulation profiles in transmen and transwomen. J Thromb Haemost. 2021 Apr;19(4):1029-1037. doi: 10.1111/jth.15256. Epub 2021 Feb 22. PMID 33527671
- [Background] Asscheman H, Gooren LJ, Eklund PL. Mortality and morbidity in transsexual patients with cross-gender hormone treatment. Metabolism. 1989 Sep;38(9):869-73. doi: 10.1016/0026-0495(89)90233-3. PMID 2528051
- [Background] Nota NM, Wiepjes CM, de Blok CJM, Gooren LJG, Kreukels BPC, den Heijer M. Occurrence of Acute Cardiovascular Events in Transgender Individuals Receiving Hormone Therapy. Circulation. 2019 Mar 12;139(11):1461-1462. doi: 10.1161/CIRCULATIONAHA.118.038584. No abstract available. PMID 30776252
- [Background] Tangpricha V, den Heijer M. Oestrogen and anti-androgen therapy for transgender women. Lancet Diabetes Endocrinol. 2017 Apr;5(4):291-300. doi: 10.1016/S2213-8587(16)30319-9. Epub 2016 Dec 2. PMID 27916515
- [Background] Eisenberger A, Westhoff C. Hormone replacement therapy and venous thromboembolism. J Steroid Biochem Mol Biol. 2014 Jul;142:76-82. doi: 10.1016/j.jsbmb.2013.08.016. Epub 2013 Sep 3. PMID 24007716
- [Background] Doll E, Gunsolus I, Thorgerson A, Tangpricha V, Lamberton N, Sarvaideo JL. Pharmacokinetics of Sublingual Versus Oral Estradiol in Transgender Women. Endocr Pract. 2022 Mar;28(3):237-242. doi: 10.1016/j.eprac.2021.11.081. Epub 2021 Nov 13. PMID 34781041
- [Background] Angus LM, Nolan BJ, Zajac JD, Cheung AS. A systematic review of antiandrogens and feminization in transgender women. Clin Endocrinol (Oxf). 2021 May;94(5):743-752. doi: 10.1111/cen.14329. Epub 2020 Oct 5. PMID 32926454
- [Background] Haupt C, Henke M, Kutschmar A, Hauser B, Baldinger S, Saenz SR, Schreiber G. Antiandrogen or estradiol treatment or both during hormone therapy in transitioning transgender women. Cochrane Database Syst Rev. 2020 Nov 28;11(11):CD013138. doi: 10.1002/14651858.CD013138.pub2. PMID 33251587
- [Background] Canonico M. Hormone therapy and risk of venous thromboembolism among postmenopausal women. Maturitas. 2015 Nov;82(3):304-7. doi: 10.1016/j.maturitas.2015.06.040. Epub 2015 Jul 26. PMID 26276103
- [Background] Peverill RE. Hormone therapy and venous thromboembolism. Best Pract Res Clin Endocrinol Metab. 2003 Mar;17(1):149-64. doi: 10.1016/s1521-690x(02)00079-9. PMID 12763518
- [Background] Yaish I, Gindis G, Greenman Y, Moshe Y, Arbiv M, Buch A, Sofer Y, Shefer G, Tordjman K. Sublingual Estradiol Offers No Apparent Advantage Over Combined Oral Estradiol and Cyproterone Acetate for Gender-Affirming Hormone Therapy of Treatment-Naive Trans Women: Results of a Prospective Pilot Study. Transgend Health. 2023 Dec 13;8(6):485-493. doi: 10.1089/trgh.2023.0022. eCollection 2023 Dec. PMID 38130980
- Available data/document: Individual Participant Data Set — https://doi.org/10.17605/OSF.IO/TCRUW